CLINICAL TRIAL: NCT04080076
Title: A Multicenter Comparative and Efficacy Study of ACTHar Gel Alone or in Combination With Tacrolimus in Fibrillary Glomerulopathy
Brief Title: Comparative and Efficacy Study of ACTHar Gel Alone or in Combination With Tacrolimus in Fibrillary Glomerulopathy
Acronym: FACT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was updated and issued a new NCT number.
Sponsor: NephroNet, Inc. (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN-
Record Dates: First submitted 2019-06-28; First posted 2019-09-06 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: ACTHar gel alone- patients will receive 80units SQ 2X/week for 52 weeks
  ACTH gel 80 units 2X per week plus oral Tacrolimus (1.0 mg BID) titrating to a trough level of 4-6 ng/ml for 52 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTHar gel combined with Tacrolimus (Active Comparator): ACTHar Gel units 2 times per week plus oral Tacrolimus (1.0 mg BID) titrating to a trough level of 4-6 ng/ml for 52 weeks
  Interventions: Drug: Acthar 80 UNT/ML Injectable Solution; Drug: Oral Tab Tacrolimus
- ACTHar gel (Active Comparator): ACTHar Gel units 2 times per week for 52 weeks
  Interventions: Drug: Acthar 80 UNT/ML Injectable Solution; Drug: Oral Tab Tacrolimus

INTERVENTIONS:
Drug: Acthar 80 UNT/ML Injectable Solution — ACTHar 80 Units SQ 1042 x Week
Drug: Oral Tab Tacrolimus — Oral Tab Tacrolimus (1.0 mg PO BID) in combination with ACTHar 80 Units SQ 2 X week

SUMMARY:
Treatment with combination ACTHar gel and Tacrolimus therapy or ACTHar gel therapy alone in lowering urinary protein to creatinine (UP/Cr) ratios

DETAILED DESCRIPTION:
This is a multicenter, Phase 4, prospective, open labeled study to compare the safety, tolerability, and efficacy of a 12month course of ACTHar Gel and Tacrolimus therapy or ACTHar gel therapy alone in lowering urinary protein to creatinine (UP/Cr) ratios.

The addition of tacrolimus patients exhiba partial to ACTH resulted in a further reduction in Fibrillary.

Spe #1-will randomize with biopsy proven DNA-JB9 positive Fibrillary glomerulopathy to receive course of ACTHar gel alone at 80 units per week or in combination with oral Tacrolimus at 1 mg BID

Hypothesis Treatment with ACTHar Gel with oral Tacrolimus will result in a higher eGFR after 24 months of follow up than patients randomized to ACTHar gel therapy alone.

Hy3: Combination therapy of ACTHar Gel and Tacrolimus in patients with DNA-JB9 positive Fibrillary will lead to significant markers of podocyte injury compared ACTHar Gel alone.

ELIGIBILITY:
Histologic Inclusion Criteria:

All patients with a diagnosis of The Fibrillary GN wbe classified according to the Nasr nomenclature:

1. Renal biopsy demonstrating JB9 Positive staining within 3 years of study randomization
2. Mesangial expansion with/without glomerular sclerosis diffuse sclerosis

4) Crescents or capillary proliferation Note: Patients with > 50% interstitial fibrosis will not be eligible for study

Inclusion Criteria:

1. Female ag
2. Biopsy proven Fibrillary GN within 3 years of study randomization
3. Stable Maximum RAAS inhibition X 40 weeks prior to randomization Note: Maximum inhibition will be the discretion of the site PI
4. eGFR > 25 mls/min
5. UP/Cr ratio > 2000 mg/gm 5 Note: IF UP/Cr less than 2000 mg/gm, a formal urine collection for total protein can be performed. The total 24-hour will need to >/= 2000mg.
6. Blood pressure targeted to < 140 at the time of randomization
7. Patients with MGUS without history of myeloma WILL be eligible.
8. Patients with monoclonal staining for fibrillary fibers will be excluded
9. Patients with Type II non-insulin dependent diabetes WILL be eligible provided the renal biopsy does not show nodular Kimmelstiel Wilson lesions

Exclusion

1. Patients with MGUS and history of myeloma WILL be eligible
2. Patients with active viral production of either B or C as evidence by historical PCR test positive for active viral shedding
3. HIV seropositivity
4. Renal biopsy data with > 5Interstitialxxxx Fibrosis
5. Patient with active or a known history
6. Patients with insulin Dependent diabetes mellitus will be excluded Note: Patients diabetes and are well controlled without the need for insulin WILL be eligible for the study.
7. Patients with Type non-insulin diabetes WILL be eligible provided the renal biopsy does not s nodular Kimmelstiel Wilson lesions.
8. Patients receiving steroids, MMF, cyc, Azathioprine or other immunosuppressive agent with of study random Note: Wash medications will be allowed at the screening visit
9. Patients having received Rituximab or cell modifying biologic bbtherapy within 60 months of randomiza

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
change in UP/Cr ratio in patients with biopsy proven Fibrillary after treated with ACTHar gel alone OR in combination with oral Tacrolimus | 12 months
  The change in UP/Cr ratio in patients with biopsy proven Fibrillary after 12 months of treatment with ACTHar gel (80 units SQ 2X/week) alone OR in combination with oral Tacrolimus (1.0 mg PO BID). The change in UP/Cr for each group will also be compared to baseline UP/Cr ratios prior to randomization

SECONDARY OUTCOMES:
relative change in UP/Cr | 24 months
  The relative change in UP/Cr at 24 months (12 months after stopping both ACTH and Tacrolimus) in the ACTHar gel group and the ACTHar gel + Tacrolimus group.
T that achieves complete, partial or clinical responses | 12 months
  The percentage of patients in the ACTHar gel alone ACTHar gel + Tacrolimus group that achieves complete, partial or clinical responses after 12 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tumlin, MD, Principal Investigator — NephroNet, Inc.
Locations (1):
- Georgia Nephrology Research Institute, Lawrenceville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Canetta P. Disentangling a Case of Glomerulonephritis with Fibrils. Clin J Am Soc Nephrol. 2022 Jul;17(7):1070-1072. doi: 10.2215/CJN.00630122. Epub 2022 Jun 2. No abstract available. PMID 35654563